CLINICAL TRIAL: NCT06004128
Title: Provide Pre-approval Single-patient Expanded Access (Compassionate Use) of VYD222 for Patients With Symptomatic COVID-19 Refractory to Other Treatments
Status: No longer available | Type: Expanded Access
Sponsor: Invivyd, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VYD222-EA-001
Record Dates: First submitted 2023-08-18; First posted 2023-08-22 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: VYD222 — Monoclonal antibody

SUMMARY:
Provide pre-approval single-patient Expanded Access (Compassionate Use) of VYD222 for patients with symptomatic COVID-19 refractory to other treatments.

Sex: All
Age Groups: Child, Adult, Older Adult